CLINICAL TRIAL: NCT05564962
Title: Quality and Independence of Gait Classification Scale for Duchenne Muscular Dystrophy (QIGS-DMD): The Development, Validity and Reliability
Brief Title: Quality and Independence of Gait Classification Scale for DMD (QIGS-DMD)
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güllü AYDIN YAĞCIOĞLU, Research Asisstant, Hacettepe University
Other Study IDs: QIGSDMD
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Duchenne Muscular Dystrophy; Gait Disorders in Children
Keywords: Duchenne Muscular Dystrophy; scale development; gait; classification; reliability; validitiy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quality and Independence of Gait Classification Scale for Duchenne Muscular Dystrophy (QIGS-DMD) — MFM is a valid and reliable measure to evaluate the severity of the motor deficit of both ambulatory and non-ambulatory children with neuromuscular diseases. MFM consists of 32 items in 3 dimensions and is scored as a percentage of the maximum possible score which higher scores indicate better functional status. VLERS is a 10-item ordinal scale that identifies the functional status of the lower limbs. According to VLERS, level 1 indicates that the patient can walk independently and climb stairs without assistance while level 10 indicates is the patient is bedridden.
  Other Names: Motor Function Measure (MFM) and Vignos Lower Extremity Rating Scale (VLERS).

SUMMARY:
The aim of this study was to develop a reliable and valid gait classification scale for Duchenne Muscular Dystrophy (QIGS-DMD). The items of the QIGS-DMD were designed based on the literature review considering existing functional classification scales, gait scales, and the opinions of the physiotherapists who were expertized in rehabilitation of patients with DMD. Content validity was determined based on the opinions of a total of ten expert physiotherapists. Videos were recorded during gait of 69 children with DMD and inter- and intra-rater reliability were examined. Criterion validity was determined according to the relationship between QIGS-DMD and Motor Function Measure (MFM) and Vignos Lower Extremity Rating Scale (VLERS).

ELIGIBILITY:
Inclusion Criteria:

* being 5 years old or above, and
* having a confirmed diagnosis of Duchenne Muscular Dystrophy.

Exclusion Criteria:

* having other coexisting medical or psychiatric diseases or injury and/or surgery related to the lower extremities within the last 6 months

Ages: 5 Years to 18 Years | Sex: Male
Age Groups: Child, Adult
Study Population: Study population consisted of patients with Duchenne Muscular Dystrophy
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Quality and Independence of Gait Classification Scale for Duchenne Muscular Dystrophy (QIGS-DMD) | 10 minutes
  It is the scale developed within the scope of the study.

SECONDARY OUTCOMES:
Motor Fucntion Measure (MFM) | 20-30 minutes
  MFM is a valid and reliable measure to evaluate the severity of the motor deficit of both ambulatory and non-ambulatory children with neuromuscular diseases. MFM consists of 32 items in 3 dimensions and is scored as a percentage of the maximum possible score which higher scores indicate better functional status.
Vignos Lower Extremity Rating Scale (VLERS) | 10 minutes
  VLERS is a 10-item ordinal scale that identifies the functional status of the lower limbs. According to VLERS, level 1 indicates that the patient can walk independently and climb stairs without assistance while level 10 indicates is the patient is bedridden

CONTACTS AND LOCATIONS:
Overall Officials: Güllü Aydın Yağcıoğlu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Güllü Aydın Yağcıoğlu, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided